CLINICAL TRIAL: NCT02632019
Title: A Clinical Study of Adoptive Cellular Immunotherapy Using Precision T Cells Specific to Personalized Neo-antigen in Treating Patients With Advanced Malignant Tumor of Biliary Tract
Brief Title: Immunotherapy Using Precision T Cells Specific to Personalized Neo-antigen for the Treatment of Advanced Malignant Tumor of Biliary Tract
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2015-02-006
Record Dates: First submitted 2015-12-12; First posted 2015-12-16 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Biliary Tract Malignant Tumor
Keywords: advanced biliary tract malignant tumor; dendritic cell; precision T cell for neo-antigen
MeSH Terms: interventions — Gemcitabine

ARMS (2):
- gemcitabine (Active Comparator): Gemcitabine treatments will be performed once a week with a total of six times
  Interventions: Drug: Gemcitabine
- Dendritic cell-precision T cell for neo-antigen (Experimental): Dendritic cell-precision T cell for neo-antigen (DC-PNAT) combined with gemcitabine treatment: Gemcitabine: once a week with a total of six times before 60 days prior to the start of drawing blood. DC-PNAT: once per 3 weeks with a total of three periods.
  Interventions: Drug: Gemcitabine; Biological: Dendritic cell-precision T cell for neo-antigen combined with gemcitabine treatment

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m2, Physiological saline 100ml:IV (in the vein) once a week with a total of six times.
Biological: Dendritic cell-precision T cell for neo-antigen combined with gemcitabine treatment — Gemcitabine: Gemcitabine 1000mg/m2, Physiological saline 100ml: IV (in the vein) once a week with a total of six times before 60 days prior to the start of drawing blood. DC-PNAT: DC cell suspension (1×107 DC+ physiological saline + 0.25% human serum albumin) 1ml for each infusion, subcutaneous injection for each infusion, 3 cycles, each cycle received two infusions on day 19, 20; 40, 41; 61, 62.
  PNAT cell suspension (1-6×109 PNAT + physiological saline + 0.25% human serum albumin) 300ml for each infusion, IV (in the vein) for each infusion, 3 cycles, each cycle received one infusions on day 21, 42, 63.
  Arms: Dendritic cell-precision T cell for neo-antigen

SUMMARY:
Objectives:

The purpose of this study is to evaluate the safety and prognosis of dendritic cell-precision T cell for neo-antigen in the treatment of advanced biliary tract malignant tumor.

Methods:

This study designs a novel therapy using dendritic cell-precision multiple antigen T cells. 40 patients will be enrolled. They are randomly divided into gemcitabine group and dendritic cell-precision T cell for neo-antigen combined with gemcitabine group. Gemcitabine treatments will be performed once a week with a total of six times. Dendritic cell-precision T cell for neo-antigen combined with gemcitabine treatment: Gemcitabine: once a week with a total of six times before 60 days prior to the start of drawing blood. Dendritic cell-precision T cell for neo-antigen: once per 3 weeks with a total of three periods. The mail clinical indicators are Progression-Free-Survival and Overall Survival.

DETAILED DESCRIPTION:
A total of 40 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18~65 years old, male or female;2. Life expectancy > 6 months;3. Eastern Cooperative Oncology Group (ECOG) score: 0-2;4. Laboratory examination: ① white blood cell ≥ 3 x 109/L. blood platelet count ≥ 60 x 109/L; hemoglobin ≥85g/L; ② total bilirubin ≤100 mol/L; aminopherase less than five times of the normal; ③ serum creatinine less than 1.5 times of the normal;5. Signed informed consent;6. Patients with fertility are willing to use contraceptive method.

Exclusion Criteria:

* 1. Expected Overall survival < 6 months;2.Other serious diseases:the heart,lung, kidney, digestive, nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, Etc.3.serum creatinine > 2.5mg/dL; Serum Glutamic Oxaloacetic Transaminase (SGOT) > 5 times of the normal;total bilirubin > 100μmol/L; 4.Other drugs, biological, chemotherapy or radiation therapy were used within 1 months;5. Without signed Informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 yeas

SECONDARY OUTCOMES:
Progress-free survival | 2 yeas
Quality of life | 2 yeas
  Quality of life core questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqing Jiang, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China

REFERENCES:
- [Background] Ilyas SI, Gores GJ. Pathogenesis, diagnosis, and management of cholangiocarcinoma. Gastroenterology. 2013 Dec;145(6):1215-29. doi: 10.1053/j.gastro.2013.10.013. Epub 2013 Oct 15. PMID 24140396
- [Background] Bergquist A, von Seth E. Epidemiology of cholangiocarcinoma. Best Pract Res Clin Gastroenterol. 2015 Apr;29(2):221-32. doi: 10.1016/j.bpg.2015.02.003. Epub 2015 Feb 16. PMID 25966423
- [Background] Cai XY, Gao Q, Qiu SJ, Ye SL, Wu ZQ, Fan J, Tang ZY. Dendritic cell infiltration and prognosis of human hepatocellular carcinoma. J Cancer Res Clin Oncol. 2006 May;132(5):293-301. doi: 10.1007/s00432-006-0075-y. Epub 2006 Jan 19. PMID 16421755
- [Background] Knippertz I, Hesse A, Schunder T, Kampgen E, Brenner MK, Schuler G, Steinkasserer A, Nettelbeck DM. Generation of human dendritic cells that simultaneously secrete IL-12 and have migratory capacity by adenoviral gene transfer of hCD40L in combination with IFN-gamma. J Immunother. 2009 Jun;32(5):524-38. doi: 10.1097/CJI.0b013e3181a28422. PMID 19609245
- [Background] Bonehill A, Van Nuffel AM, Corthals J, Tuyaerts S, Heirman C, Francois V, Colau D, van der Bruggen P, Neyns B, Thielemans K. Single-step antigen loading and activation of dendritic cells by mRNA electroporation for the purpose of therapeutic vaccination in melanoma patients. Clin Cancer Res. 2009 May 15;15(10):3366-75. doi: 10.1158/1078-0432.CCR-08-2982. Epub 2009 May 5. PMID 19417017
- [Background] Bellik L, Gerlini G, Parenti A, Ledda F, Pimpinelli N, Neri B, Pantalone D. Role of conventional treatments on circulating and monocyte-derived dendritic cells in colorectal cancer. Clin Immunol. 2006 Oct;121(1):74-80. doi: 10.1016/j.clim.2006.06.011. Epub 2006 Aug 17. PMID 16914380
- [Background] Babatz J, Rollig C, Lobel B, Folprecht G, Haack M, Gunther H, Kohne CH, Ehninger G, Schmitz M, Bornhauser M. Induction of cellular immune responses against carcinoembryonic antigen in patients with metastatic tumors after vaccination with altered peptide ligand-loaded dendritic cells. Cancer Immunol Immunother. 2006 Mar;55(3):268-76. doi: 10.1007/s00262-005-0021-x. Epub 2005 Jul 21. PMID 16034561
- [Background] Fay JW, Palucka AK, Paczesny S, Dhodapkar M, Johnston DA, Burkeholder S, Ueno H, Banchereau J. Long-term outcomes in patients with metastatic melanoma vaccinated with melanoma peptide-pulsed CD34(+) progenitor-derived dendritic cells. Cancer Immunol Immunother. 2006 Oct;55(10):1209-18. doi: 10.1007/s00262-005-0106-6. Epub 2005 Dec 6. PMID 16331519
- [Background] Davis ID, Chen Q, Morris L, Quirk J, Stanley M, Tavarnesi ML, Parente P, Cavicchiolo T, Hopkins W, Jackson H, Dimopoulos N, Tai TY, MacGregor D, Browning J, Svobodova S, Caron D, Maraskovsky E, Old LJ, Chen W, Cebon J. Blood dendritic cells generated with Flt3 ligand and CD40 ligand prime CD8+ T cells efficiently in cancer patients. J Immunother. 2006 Sep-Oct;29(5):499-511. doi: 10.1097/01.cji.0000211299.29632.8c. PMID 16971806
- [Background] Escobar A, Lopez M, Serrano A, Ramirez M, Perez C, Aguirre A, Gonzalez R, Alfaro J, Larrondo M, Fodor M, Ferrada C, Salazar-Onfray F. Dendritic cell immunizations alone or combined with low doses of interleukin-2 induce specific immune responses in melanoma patients. Clin Exp Immunol. 2005 Dec;142(3):555-68. doi: 10.1111/j.1365-2249.2005.02948.x. PMID 16297169
- [Background] Thomas-Kaskel AK, Zeiser R, Jochim R, Robbel C, Schultze-Seemann W, Waller CF, Veelken H. Vaccination of advanced prostate cancer patients with PSCA and PSA peptide-loaded dendritic cells induces DTH responses that correlate with superior overall survival. Int J Cancer. 2006 Nov 15;119(10):2428-34. doi: 10.1002/ijc.22097. PMID 16977630
- [Background] Fuessel S, Meye A, Schmitz M, Zastrow S, Linne C, Richter K, Lobel B, Hakenberg OW, Hoelig K, Rieber EP, Wirth MP. Vaccination of hormone-refractory prostate cancer patients with peptide cocktail-loaded dendritic cells: results of a phase I clinical trial. Prostate. 2006 Jun 1;66(8):811-21. doi: 10.1002/pros.20404. PMID 16482569
- [Background] Kyte JA, Gaudernack G. Immuno-gene therapy of cancer with tumour-mRNA transfected dendritic cells. Cancer Immunol Immunother. 2006 Nov;55(11):1432-42. doi: 10.1007/s00262-006-0161-7. Epub 2006 Apr 13. PMID 16612595
- [Background] Wang QJ, Hanada K, Perry-Lalley D, Bettinotti MP, Karpova T, Khong HT, Yang JC. Generating renal cancer-reactive T cells using dendritic cells (DCs) to present autologous tumor. J Immunother. 2005 Nov-Dec;28(6):551-9. doi: 10.1097/01.cji.0000175495.13476.1f. PMID 16224272
- [Background] Holtl L, Ramoner R, Zelle-Rieser C, Gander H, Putz T, Papesh C, Nussbaumer W, Falkensammer C, Bartsch G, Thurnher M. Allogeneic dendritic cell vaccination against metastatic renal cell carcinoma with or without cyclophosphamide. Cancer Immunol Immunother. 2005 Jul;54(7):663-70. doi: 10.1007/s00262-004-0629-2. Epub 2004 Dec 17. PMID 15918076
- [Background] Ferrari S, Malugani F, Rovati B, Porta C, Riccardi A, Danova M. Flow cytometric analysis of circulating dendritic cell subsets and intracellular cytokine production in advanced breast cancer patients. Oncol Rep. 2005 Jul;14(1):113-20. PMID 15944777
- [Background] Bohnenkamp HR, Coleman J, Burchell JM, Taylor-Papadimitriou J, Noll T. Breast carcinoma cell lysate-pulsed dendritic cells cross-prime MUC1-specific CD8+ T cells identified by peptide-MHC-class-I tetramers. Cell Immunol. 2004 Sep-Oct;231(1-2):112-25. doi: 10.1016/j.cellimm.2004.12.007. Epub 2005 Feb 8. PMID 15919376
- [Background] Chen W, Chan AS, Dawson AJ, Liang X, Blazar BR, Miller JS. FLT3 ligand administration after hematopoietic cell transplantation increases circulating dendritic cell precursors that can be activated by CpG oligodeoxynucleotides to enhance T-cell and natural killer cell function. Biol Blood Marrow Transplant. 2005 Jan;11(1):23-34. doi: 10.1016/j.bbmt.2004.08.004. PMID 15625541
- [Background] Triozzi PL, Khurram R, Aldrich WA, Walker MJ, Kim JA, Jaynes S. Intratumoral injection of dendritic cells derived in vitro in patients with metastatic cancer. Cancer. 2000 Dec 15;89(12):2646-54. doi: 10.1002/1097-0142(20001215)89:123.0.co;2-a. PMID 11135227
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Gubin MM, Zhang X, Schuster H, Caron E, Ward JP, Noguchi T, Ivanova Y, Hundal J, Arthur CD, Krebber WJ, Mulder GE, Toebes M, Vesely MD, Lam SS, Korman AJ, Allison JP, Freeman GJ, Sharpe AH, Pearce EL, Schumacher TN, Aebersold R, Rammensee HG, Melief CJ, Mardis ER, Gillanders WE, Artyomov MN, Schreiber RD. Checkpoint blockade cancer immunotherapy targets tumour-specific mutant antigens. Nature. 2014 Nov 27;515(7528):577-81. doi: 10.1038/nature13988. PMID 25428507
- [Background] Yadav M, Jhunjhunwala S, Phung QT, Lupardus P, Tanguay J, Bumbaca S, Franci C, Cheung TK, Fritsche J, Weinschenk T, Modrusan Z, Mellman I, Lill JR, Delamarre L. Predicting immunogenic tumour mutations by combining mass spectrometry and exome sequencing. Nature. 2014 Nov 27;515(7528):572-6. doi: 10.1038/nature14001. PMID 25428506
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015 Apr 3;348(6230):56-61. doi: 10.1126/science.aaa8172. PMID 25838373
- [Background] Fischbach MA, Bluestone JA, Lim WA. Cell-based therapeutics: the next pillar of medicine. Sci Transl Med. 2013 Apr 3;5(179):179ps7. doi: 10.1126/scitranslmed.3005568. PMID 23552369
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Background] Robbins PF, Lu YC, El-Gamil M, Li YF, Gross C, Gartner J, Lin JC, Teer JK, Cliften P, Tycksen E, Samuels Y, Rosenberg SA. Mining exomic sequencing data to identify mutated antigens recognized by adoptively transferred tumor-reactive T cells. Nat Med. 2013 Jun;19(6):747-52. doi: 10.1038/nm.3161. Epub 2013 May 5. PMID 23644516
- [Background] Tran E, Turcotte S, Gros A, Robbins PF, Lu YC, Dudley ME, Wunderlich JR, Somerville RP, Hogan K, Hinrichs CS, Parkhurst MR, Yang JC, Rosenberg SA. Cancer immunotherapy based on mutation-specific CD4+ T cells in a patient with epithelial cancer. Science. 2014 May 9;344(6184):641-5. doi: 10.1126/science.1251102. PMID 24812403
- [Background] Curtsinger JM, Mescher MF. Inflammatory cytokines as a third signal for T cell activation. Curr Opin Immunol. 2010 Jun;22(3):333-40. doi: 10.1016/j.coi.2010.02.013. Epub 2010 Apr 2. PMID 20363604
- [Background] Zinkernagel RM, Doherty PC. Restriction of in vitro T cell-mediated cytotoxicity in lymphocytic choriomeningitis within a syngeneic or semiallogeneic system. Nature. 1974 Apr 19;248(5450):701-2. doi: 10.1038/248701a0. No abstract available. PMID 4133807
- [Background] Lafferty KJ, Warren HS, Woolnough JA. A mediator acting as a costimulator for the development of cytotoxic responses in vitro. Adv Exp Med Biol. 1979;114:497-501. doi: 10.1007/978-1-4615-9101-6_82. No abstract available. PMID 313677
- [Background] Turtle CJ, Hudecek M, Jensen MC, Riddell SR. Engineered T cells for anti-cancer therapy. Curr Opin Immunol. 2012 Oct;24(5):633-9. doi: 10.1016/j.coi.2012.06.004. Epub 2012 Jul 18. PMID 22818942
- [Background] Morgan RA, Dudley ME, Wunderlich JR, Hughes MS, Yang JC, Sherry RM, Royal RE, Topalian SL, Kammula US, Restifo NP, Zheng Z, Nahvi A, de Vries CR, Rogers-Freezer LJ, Mavroukakis SA, Rosenberg SA. Cancer regression in patients after transfer of genetically engineered lymphocytes. Science. 2006 Oct 6;314(5796):126-9. doi: 10.1126/science.1129003. Epub 2006 Aug 31. PMID 16946036
- [Background] Santarpia M, Karachaliou N. Tumor immune microenvironment characterization and response to anti-PD-1 therapy. Cancer Biol Med. 2015 Jun;12(2):74-8. doi: 10.7497/j.issn.2095-3941.2015.0022. No abstract available. PMID 26175922
- [Background] Nagaraj S, Gabrilovich DI. Tumor escape mechanism governed by myeloid-derived suppressor cells. Cancer Res. 2008 Apr 15;68(8):2561-3. doi: 10.1158/0008-5472.CAN-07-6229. PMID 18413722
- [Background] Staveley-O'Carroll K, Sotomayor E, Montgomery J, Borrello I, Hwang L, Fein S, Pardoll D, Levitsky H. Induction of antigen-specific T cell anergy: An early event in the course of tumor progression. Proc Natl Acad Sci U S A. 1998 Feb 3;95(3):1178-83. doi: 10.1073/pnas.95.3.1178. PMID 9448305
- [Background] Boon T, Coulie PG, Van den Eynde BJ, van der Bruggen P. Human T cell responses against melanoma. Annu Rev Immunol. 2006;24:175-208. doi: 10.1146/annurev.immunol.24.021605.090733. PMID 16551247
- [Background] Lee PP, Yee C, Savage PA, Fong L, Brockstedt D, Weber JS, Johnson D, Swetter S, Thompson J, Greenberg PD, Roederer M, Davis MM. Characterization of circulating T cells specific for tumor-associated antigens in melanoma patients. Nat Med. 1999 Jun;5(6):677-85. doi: 10.1038/9525. PMID 10371507
- [Background] Radoja S, Saio M, Frey AB. CD8+ tumor-infiltrating lymphocytes are primed for Fas-mediated activation-induced cell death but are not apoptotic in situ. J Immunol. 2001 May 15;166(10):6074-83. doi: 10.4049/jimmunol.166.10.6074. PMID 11342625
- [Background] Radoja S, Saio M, Schaer D, Koneru M, Vukmanovic S, Frey AB. CD8(+) tumor-infiltrating T cells are deficient in perforin-mediated cytolytic activity due to defective microtubule-organizing center mobilization and lytic granule exocytosis. J Immunol. 2001 Nov 1;167(9):5042-51. doi: 10.4049/jimmunol.167.9.5042. PMID 11673513
- [Background] Driessens G, Kline J, Gajewski TF. Costimulatory and coinhibitory receptors in anti-tumor immunity. Immunol Rev. 2009 May;229(1):126-44. doi: 10.1111/j.1600-065X.2009.00771.x. PMID 19426219